CLINICAL TRIAL: NCT04189991
Title: Oxygen Titration Protocol for Exertion of COPD Patients by an Automated Adjustment Device: a Monocentric, Prospective, Cross-over Study.
Brief Title: Oxygen Titration Protocol for Exertion of COPD Patients by an Automated Adjustment Device
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has not started yet due to COVID pandemic.
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Osixeno
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: COPD; Chronic Respiratory Insufficiency
Keywords: COPD; Long-term oxygen therapy; Six minutes walk test; Exertion; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients will undergo titration 6 minutes walk test using the standard and the automatic method in random order.
Who Masked: Participant
Masking Description: The same device will be used for both oxygen titration protocol and during 6 minutes walk tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual then automated oxygen titration (Active Comparator): First will be performed the manual oxygen titration and then the automatic oxygen titration.
  Interventions: Device: Free 02
- Automatic then manual oxygen titration (Active Comparator): First will be performed the automatic oxygen titration and then the manual oxygen titration.
  Interventions: Device: Free 02

INTERVENTIONS:
Device: Free 02 — With the manual oxygen titration, the physiotherapist adjust manually the oxygen flow using the FreeO2 device during a titration 6 minutes walk test.
  With the automated adjustment oxygen titration, the flow will be self adjusted by the FreeO2 device during a titration 6 minutes walk test. In that hase, the median flow rate and the 95th flow rate will be evaluated during the validation 6 minutes walk test.

SUMMARY:
The aim of our study is to assess if an automated titration of oxygen flow during exertion can be a useful tool to determinate the level of oxygen required by COPD patients that are using oxygen therapy during exercise.

DETAILED DESCRIPTION:
All patients referred to our centre of oxygen titration during exertion will be offered to participate in our study.

After baseline assessments, patients will have an oxygen titration using two different methods in random order:

* Usual titration protocol will include an manual oxygen increase during a titration 6 minutes walk test
* Automatic titration protocol that will use the automated oxygen titration device to adjust oxygen flow rate during a titration 6 minutes walk test.

After each titration protocol, the efficacy of the titration will be assessed in 3 validation 6 minutes walk tests during which oxygen flow will be set at:

* The manually determined flow rate
* The 95th percentile flow rate of the automatic titration
* The median flow rate of the automatic titration

During validation 6 minutes walk test, oxygen saturation, dyspnea, walked distance and heart rate will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 85 years
* COPD patients at the stage of CRF under LTOT or desaturating at exercise
* Written and signed consent

Exclusion Criteria:

* Patients under guardianship or curatorship.
* Pregnant women
* Patients with non-weaned smoking.
* Patients using technical assistance to move
* Inability to perform 6MWT due to locomotor disorders.
* Inability to understand 6MWT due to cognitive disorders
* Patients exacerbating
* Unstable angora
* myocardial infarction < 1 month
* HR at rest > 120 bpm
* systolic blood pressure > 18 and/or diastolic blood pressure > 10

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time spent in the pulse oxygen saturation target (Sp02) which is 92% +/- 2 during validation 6 minutes walk-test | 6 minutes
  The time spent will be retrieved from the oxygen delivery device. it will be expressed in percentage of time of the 6 minutes walk tests and seconds.

SECONDARY OUTCOMES:
Time spent with "moderate hypoxemia" (Sp02 <90%), "severe hypoxemia" (Sp02 <85%) or "hyperoxia" (Sp02> 94%). | 6 minutes
  The time spent will be retrieved from the oxygen delivery device. it will be expressed in percentage of time of the 6 minutes walk tests and seconds.

OTHER OUTCOMES:
Oxygen saturation | Before, after the 6MWT, 1 minute after the end of the 6MWT, 3 minutes, 6 minutes, 10 minutes.
  The oxygen saturation will be retrieved from the oxygen delivery device. it will be expressed in percentage of time of the 6 minutes walk tests and seconds.
Heart rate | Before, after the 6MWT, 1 minute after the end of the 6MWT, 3 minutes, 6 minutes, 10 minutes.
  The heart rate will be retrieved from the oxygen delivery device. it will be expressed in percentage of time of the 6 minutes walk tests and seconds.
Dyspnoea | Before, after the 6MWT, 1 minute after the end of the 6MWT, 3 minutes, 6 minutes, 10 minutes.
  The dyspnea will be assessed using a BORG scale (0: Rest to 10: Maximal)
Tiredness of the lower limbs | Before, after the 6MWT, 1 minute after the end of the 6MWT, 3 minutes, 6 minutes, 10 minutes.
  Tiredness of the lower limbs will be assessed using a visual analogue scale (0: No tiredness at all to 10: Maximal tiredness)
Distance walked during the validation 6 minutes walk test | 6 minutes
  THe distance will be measured using a metered corridor with a meter precision
Time spent to perform the titrations | 30 minutes
  The time spent for each titration procedure will be assessed using a chronometer.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Patout, MD, Study Chair — ADIR Association; Antoine Cuvelier, PhD, Principal Investigator — ADIR Association; Jean-François Muir, PhD, Study Chair — ADIR Association; Pauline Smondack, PT, Study Chair — ADIR Association
Locations (1):
- CHU Charles Nicolle, Rouen, France

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data from the trial will be available upon reasonnable request to the corresponding author. Data will not be made available for any commercial use.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After study completion and for 10 years.
Access Criteria: Researchers

REFERENCES:
- [Background] Bon usage des technologies de santé, HAS, Oxygénothérapie à long terme : choisir la source la mieux adaptée, Mai 2012.
- [Background] Journal Officiel de la République Française, Arrêté du 23 février 2015, Oxygénothérapie, Février 2015.
- [Background] Kim V, Benditt JO, Wise RA, Sharafkhaneh A. Oxygen therapy in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2008 May 1;5(4):513-8. doi: 10.1513/pats.200708-124ET. PMID 18453364
- [Background] Delample D, Sabate M, Prefaut C, Durand F. Does prior training affect acute O(2) supply responses during exercise in Desaturator COPD patients? Open Respir Med J. 2008;2:29-34. doi: 10.2174/1874306400802010029. Epub 2008 Mar 13. PMID 19340322
- [Background] Galera R, Casitas R, Martinez E, Lores V, Rojo B, Carpio C, Llontop C, Garcia-Rio F. Exercise oxygen flow titration methods in COPD patients with respiratory failure. Respir Med. 2012 Nov;106(11):1544-50. doi: 10.1016/j.rmed.2012.06.021. Epub 2012 Jul 21. PMID 22819520
- [Background] Ora J, Calzetta L, Pezzuto G, Senis L, Paone G, Mari A, Portalone S, Rogliani P, Puxeddu E, Saltini C. A 6MWT index to predict O2 flow correcting exercise induced SpO2 desaturation in ILD. Respir Med. 2013 Dec;107(12):2014-21. doi: 10.1016/j.rmed.2013.10.002. Epub 2013 Oct 10. PMID 24161677
- [Background] Lellouche F, L'her E. Automated oxygen flow titration to maintain constant oxygenation. Respir Care. 2012 Aug;57(8):1254-62. doi: 10.4187/respcare.01343. Epub 2012 Feb 17. PMID 22348812
- [Background] Lellouche F, Bouchard PA, Roberge M, Simard S, L'Her E, Maltais F, Lacasse Y. Automated oxygen titration and weaning with FreeO2 in patients with acute exacerbation of COPD: a pilot randomized trial. Int J Chron Obstruct Pulmon Dis. 2016 Aug 24;11:1983-90. doi: 10.2147/COPD.S112820. eCollection 2016. PMID 27601891
- [Background] Cirio S, Nava S. Pilot study of a new device to titrate oxygen flow in hypoxic patients on long-term oxygen therapy. Respir Care. 2011 Apr;56(4):429-34. doi: 10.4187/respcare.00983. Epub 2011 Jan 21. PMID 21255511
- [Background] Lellouche F, L'Her E, Bouchard PA, Brouillard C, Maltais F. Automatic Oxygen Titration During Walking in Subjects With COPD: A Randomized Crossover Controlled Study. Respir Care. 2016 Nov;61(11):1456-1464. doi: 10.4187/respcare.04406. Epub 2016 Oct 18. PMID 27794080
- [Background] Vivodtzev I, L'Her E, Vottero G, Yankoff C, Tamisier R, Maltais F, Lellouche F, Pepin JL. Automated O2 titration improves exercise capacity in patients with hypercapnic chronic obstructive pulmonary disease: a randomised controlled cross-over trial. Thorax. 2019 Mar;74(3):298-301. doi: 10.1136/thoraxjnl-2018-211967. Epub 2018 Aug 30. PMID 30166425
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- See also: Commercial description of the device used in the trial — https://www.oxynov.com/freeo2/